CLINICAL TRIAL: NCT02224196
Title: Comparison of Peak Airway Pressure and Gastric Insufflation in Manual Ventilation and Pressure-controlled Ventilation With Facemask During Anesthesia Induction in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 4-2014-0270
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Elective Urologic Surgeries
Keywords: manual ventilation; pressure-controlled ventilation; peak airway pressure; antral area

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- manual ventilation (Experimental)
  Interventions: Other: manual ventilation
- pressure-controlled ventilation (Active Comparator)
  Interventions: Other: pressure-controlled ventilation

INTERVENTIONS:
Other: manual ventilation — Anesthesia will be induced by propofol 1mg/kg via intravenous line. Once loss of eyelash reflex occurred, ultrasonography of antral area will be started by same physician. After administration of muscle relaxant (rocuronium 0.2-0.4mg/kg), manual ventilation will be performed with respiratory rate 20 breathes/min, I:E ratio of 1:1 and tidal volume with 9-10mL/kg. The pop-off valve will be set at 15cmH2O at fixed gas flow of 500mL/min of oxygen. Pressure-controlled ventilation will be performed with respiratory rate 20 breaths/min, I:E ratio of 1:1 and peak airway pressure will be set to get a tidal volume of 9-10mL/kg. The peak airway pressure during facemask ventilation will be checked. Another physician will auscultate the epigastric area to detect gastric insufflation during facemask ventilation. Ultrasonography of antral area will be checked once again after 3 minutes of facemask ventilation.
  Arms: manual ventilation
Other: pressure-controlled ventilation — Anesthesia will be induced by propofol 1mg/kg via intravenous line. Once loss of eyelash reflex occurred, ultrasonography of antral area will be started by same physician. After administration of muscle relaxant (rocuronium 0.2-0.4mg/kg), manual ventilation will be performed with respiratory rate 20 breathes/min, I:E ratio of 1:1 and tidal volume with 9-10mL/kg. The pop-off valve will be set at 15cmH2O at fixed gas flow of 500mL/min of oxygen. Pressure-controlled ventilation will be performed with respiratory rate 20 breaths/min, I:E ratio of 1:1 and peak airway pressure will be set to get a tidal volume of 9-10mL/kg. The peak airway pressure during facemask ventilation will be checked. Another physician will auscultate the epigastric area to detect gastric insufflation during facemask ventilation. Ultrasonography of antral area will be checked once again after 3 minutes of facemask ventilation.
  Arms: pressure-controlled ventilation

SUMMARY:
Comparison of peak airway pressure and gastric insufflation in manual ventilation and pressure-controlled ventilation with facemask during anesthesia induction in children.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status with I or II
2. Those parents who signed with informed consents.
3. Children who are scheduled for elective urologic surgery (aged 6 month to 7 year)

Exclusion Criteria:

1. Risk of aspiration
2. Oropharyngeal or facial anomaly
3. history of abdominal (stomach) surgery

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
peak airway pressure | 3 minutes
  The primary outcome is the difference of peak airway pressure produced by manual ventilation group and pressure-controlled ventilation group during induction of anesthesia.

SECONDARY OUTCOMES:
antral area of stomach | 3 minutes
  All patients' antral area of stomach will be calculated by ultrasound after 3 minutes-facemask ventilation to estimate the quantity of gas insufflation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Pain Medicine, Yonsei university college of medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Result] von Goedecke A, Voelckel WG, Wenzel V, Hormann C, Wagner-Berger HG, Dorges V, Lindner KH, Keller C. Mechanical versus manual ventilation via a face mask during the induction of anesthesia: a prospective, randomized, crossover study. Anesth Analg. 2004 Jan;98(1):260-263. doi: 10.1213/01.ANE.0000096190.36875.67. PMID 14693633
- [Result] Kluger MT, Visvanathan T, Myburgh JA, Westhorpe RN. Crisis management during anaesthesia: regurgitation, vomiting, and aspiration. Qual Saf Health Care. 2005 Jun;14(3):e4. doi: 10.1136/qshc.2002.004259. PMID 15933301
- [Result] Neelakanta G, Chikyarappa A. A review of patients with pulmonary aspiration of gastric contents during anesthesia reported to the Departmental Quality Assurance Committee. J Clin Anesth. 2006 Mar;18(2):102-7. doi: 10.1016/j.jclinane.2005.07.002. PMID 16563326
- [Result] Borland LM, Sereika SM, Woelfel SK, Saitz EW, Carrillo PA, Lupin JL, Motoyama EK. Pulmonary aspiration in pediatric patients during general anesthesia: incidence and outcome. J Clin Anesth. 1998 Mar;10(2):95-102. doi: 10.1016/s0952-8180(97)00250-x. PMID 9524892
- [Result] Weiler N, Latorre F, Eberle B, Goedecke R, Heinrichs W. Respiratory mechanics, gastric insufflation pressure, and air leakage of the laryngeal mask airway. Anesth Analg. 1997 May;84(5):1025-8. doi: 10.1097/00000539-199705000-00013. PMID 9141925
- [Result] Weiler N, Heinrichs W, Dick W. Assessment of pulmonary mechanics and gastric inflation pressure during mask ventilation. Prehosp Disaster Med. 1995 Apr-Jun;10(2):101-5. doi: 10.1017/s1049023x00041807. PMID 10155411
- [Result] Seet MM, Soliman KM, Sbeih ZF. Comparison of three modes of positive pressure mask ventilation during induction of anaesthesia: a prospective, randomized, crossover study. Eur J Anaesthesiol. 2009 Nov;26(11):913-6. doi: 10.1097/EJA.0b013e328329b0ab. PMID 19390448
- [Result] Ho-Tai LM, Devitt JH, Noel AG, O'Donnell MP. Gas leak and gastric insufflation during controlled ventilation: face mask versus laryngeal mask airway. Can J Anaesth. 1998 Mar;45(3):206-11. doi: 10.1007/BF03012903. PMID 9579256
- [Result] SNOW RG. THE MUSCLE RELAXANTS AND THE CARDIA, INCLUDING THE CLINICAL MANAGEMENT OF PATIENTS LIKELY TO VOMIT AND REGURGITATE. Br J Anaesth. 1963 Sep;35:541-5. doi: 10.1093/bja/35.9.541. No abstract available. PMID 14066104
- [Result] Lawes EG, Campbell I, Mercer D. Inflation pressure, gastric insufflation and rapid sequence induction. Br J Anaesth. 1987 Mar;59(3):315-8. doi: 10.1093/bja/59.3.315. PMID 3828180
- [Result] Lagarde S, Semjen F, Nouette-Gaulain K, Masson F, Bordes M, Meymat Y, Cros AM. Facemask pressure-controlled ventilation in children: what is the pressure limit? Anesth Analg. 2010 Jun 1;110(6):1676-9. doi: 10.1213/ANE.0b013e3181d8a14c. Epub 2010 Apr 30. PMID 20435941
- [Result] Moynihan RJ, Brock-Utne JG, Archer JH, Feld LH, Kreitzman TR. The effect of cricoid pressure on preventing gastric insufflation in infants and children. Anesthesiology. 1993 Apr;78(4):652-6. doi: 10.1097/00000542-199304000-00007. PMID 8466065
- [Result] Bouvet L, Albert ML, Augris C, Boselli E, Ecochard R, Rabilloud M, Chassard D, Allaouchiche B. Real-time detection of gastric insufflation related to facemask pressure-controlled ventilation using ultrasonography of the antrum and epigastric auscultation in nonparalyzed patients: a prospective, randomized, double-blind study. Anesthesiology. 2014 Feb;120(2):326-34. doi: 10.1097/ALN.0000000000000094. PMID 24317204
- [Result] Bouvet L, Mazoit JX, Chassard D, Allaouchiche B, Boselli E, Benhamou D. Clinical assessment of the ultrasonographic measurement of antral area for estimating preoperative gastric content and volume. Anesthesiology. 2011 May;114(5):1086-92. doi: 10.1097/ALN.0b013e31820dee48. PMID 21364462
- [Result] Schmitz A, Thomas S, Melanie F, Rabia L, Klaghofer R, Weiss M, Kellenberger C. Ultrasonographic gastric antral area and gastric contents volume in children. Paediatr Anaesth. 2012 Feb;22(2):144-9. doi: 10.1111/j.1460-9592.2011.03718.x. Epub 2011 Oct 14. PMID 21999211
- [Result] Brimacomb J, Keller C, Kurian S, Myles J. Reliability of epigastric auscultation to detect gastric insufflation. Br J Anaesth. 2002 Jan;88(1):127-9. doi: 10.1093/bja/88.1.127. PMID 11881867